CLINICAL TRIAL: NCT06187610
Title: Digital Intervention for Gastrointestinal (GI) Cancer Patients: A Case Study on Enhancing Symptom Self-Management During Treatment
Brief Title: Digital Delivery of Patient Education: A Case Study of Symptom Self-Management During Cancer Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel Aviv University (Other)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Principal Investigator, Ilana Dubovi, Principal Investigator, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CancerEducationTau
Record Dates: First submitted 2023-12-17; First posted 2024-01-02 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Digital Education Interventions; Knowledge Types (Mechanistic Versus Procedural)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational intervention group (Experimental)
  Interventions: Behavioral: Digital education
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Digital education — Patients assigned to the experimental group will learn about symptom self-management in a digital learning environment.
  Arms: Educational intervention group

SUMMARY:
The increasing shift from face-to-face to online patient-clinician encounters in the healthcare system requires patients to be more involved in their medical care. This raises the urgent need to evaluate the extent to which proactive patients' self-care can be supported, particularly by informed telemedicine digital channels. Despite this imperative, research offering evidence-based instructional design of digital education remains surprisingly scarce. Embracing the framework of science education, which highlights the functional role of different knowledge types in educational processes, the current study seeks to evaluate an educational approach aimed at supporting cancer patients undergoing chemotherapy.

Cancer treatment serves as an exemplar health condition, demanding daily self-management from patients. The objectives of our research are as follows: (1) To delineate the types of knowledge required for effective symptom management, active participation in one's healthcare, and judicious decision-making regarding emergency room (ER) visits, with a focus on mechanistic knowledge pertaining to the rationale for treatment and procedural knowledge concerning the treatment regimen. (2) To appraise the impact of a digital learning environment in contrast to traditional methods on patients' acquisition of mechanistic and procedural knowledge. (3) To identify how patients engage with the digital patient education environment aiming to outline leaning patterns.

The investigators hypothesize that implementing digital education will enhance patients' understanding of both the 'why' (mechanistic) and 'how' (procedural) aspects of their treatment. Importantly, the investigators expect that mechanistic knowledge will be more impactful than procedural knowledge, leading to better symptom management and patient involvement, and ultimately reducing unnecessary visits to the ER.

ELIGIBILITY:
Inclusion Criteria:

* Gastrointestinal (GI) cancer patients
* Chemotherapy session within a specific round of treatment, with eligible treatments including FOLFOX, FOLFIRINOX, and FLOT.
* Hebrew speakers.

Exclusion Criteria:

* Impaired or degraded cognitive capabilities that may hinder effective learning.
* Individuals who discontinue their treatments due to terminal advancement of their disease or death.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Symptom self-management knowledge | The test will be conducted in two time-points of the study, Time 0 (pre) and Time 2 (after two months)
  Measured by performance accuracy in a cancer-specific knowledge test

SECONDARY OUTCOMES:
Self-efficacy in symptom management | The questionnaire will be administered three times: Time 0 (pre) and Time 2 (after two months)
  Measured by self-report Self-Efficacy for Managing Chronic Disease 6-Item Scale. The scale ranges from 1 (not confident) to 10 (very confident). A higher score is interpreted as a better self-efficacy.
Confidence in decision making | The questionnaire will be administered in two time-points of the study, Time 0 (pre) and Time 2 (after two months)
  Measured by the self-report Decision Self-Efficacy Scale, which assesses patients' self-confidence in their ability to make decisions. It includes 11 items on a scale ranging from 0 (not at all confident) to 4 (very confident). A higher score is interpreted as higher confidence.
Patients engagement while learning | on Time 2, namely about two weeks to four weeks after recruitment
  Patients engagement with patient education material will be captured by psychophysiological parameters of eye-tracking and facial expressions

CONTACTS AND LOCATIONS:
Locations (1):
- Ichilov Hospital, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
upon request